CLINICAL TRIAL: NCT02081898
Title: Three-year Mild Calorie Restriction Partially Protects Against Age-related Increase in Sphingomyelin and Reduces Obesity-associated Amino Acids
Brief Title: Effects of Long Term Calorie Restriction on Sphingomyelin and Amino Acids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: wt loss_20140305
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Overweight; Obese
Keywords: low calorie diet; BMI; sphingomyelin; L-leucine; L-phenylalanine
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet, Reducing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): weight maintenance diet
- low calorie diet (LCD) group (Experimental): approximate 100 kcal/d calorie deficit
  Interventions: Dietary Supplement: LCD

INTERVENTIONS:
Dietary Supplement: LCD — approximate 100 kcal/d caloric deficit
  Other Names: weight loss diet
  Arms: low calorie diet (LCD) group

SUMMARY:
The effect of weight loss with long-term low calorie diet (LCD) on plasma metabolites is unknown. The aim was to examine whether a LCD-induced weight reduction results in changes in the extended plasma metabolites.

DETAILED DESCRIPTION:
Overweight/obese subjects (25≤ BMI <33 kg/m2) aged 40 to 59 years consumed a LCD (an approximate 100 kcal/day calorie deficit) or a weight-maintenance diet (control) in a randomized, controlled design with 3-year intervention period.

ELIGIBILITY:
Inclusion Criteria:

* 25 <= BMI < 33 kg/m2

Exclusion Criteria:

* type 2 diabetes
* cardiovascular disease
* psychiatric problems
* any medication use

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
anthropometry | 3-year follow-up
  weight, height, BMI, waist circumference, blood pressure

SECONDARY OUTCOMES:
biochemistry analysis | 3-year follow-up
  total-cholesterol, LDL-cholesterol, HDL-cholesterol, triglyceride, free fatty acids, glucose, insulin, HOMA-IR, Lp-PLA2

OTHER OUTCOMES:
plasma metabolites | 3-year follow-up
  palmitic amide, oleamide, lysoPC (16:1, 16:0, 17:0, 18:2, 18:1, 18:0, 20:4, 20:3, 22:6), PC (16:0/20:5, 16:0/20:5, 18:2/18:2, 18:0/20:4), lactosylceramide (d18:1/12:2)

CONTACTS AND LOCATIONS:
Overall Officials: Minjoo Kim, MS, Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Seoul, South Korea

REFERENCES:
- [Derived] Kim M, Lee SH, Lee JH. Global Metabolic Profiling of Plasma Shows that Three-Year Mild-Caloric Restriction Lessens an Age-Related Increase in Sphingomyelin and Reduces L-leucine and L-phenylalanine in Overweight and Obese Subjects. Aging Dis. 2016 Dec 1;7(6):721-733. doi: 10.14336/AD.2016.0330. eCollection 2016 Dec. PMID 28053823